# **Research Title**

The effect of a comprehensive dementia education program on improving attitudes toward people living with dementia: a Randomized Controlled Trial



**NCT** number:

**Document date: 2025/11/16** 

UNIVERSITAS AIRLANGGA

November, 2025

### Clinical Trial

## 1. Study Overview

Title: The Effect of a Comprehensive Dementia Education Program on Improving Attitudes

Toward People Living with Dementia: A Randomized Controlled Trial

Acronym: VReducationRCT Sponsor: Universitas Airlangga

Version: 1.0

Date: November 2025

## 2. Background and Rationale

Dementia education is critical for preparing future nurses to care for an aging population. VR-based educational programs have shown promise in improving empathy, knowledge, and attitudes. This study tests a VR dementia education program among Indonesian nursing students using an RCT design.

# 3. Study Objectives

Primary Objective:

To evaluate the effect of a comprehensive VR dementia education program on attitudes toward people living with dementia.

## Secondary Objectives:

- To measure changes in dementia knowledge.
- To assess intention to help persons living with dementia.
- To evaluate user experience and satisfaction with the VR program.

### 4. Study Design

Design: Parallel-group, open-label RCT.

Arms:

Experimental: VR Dementia Education Program
 Active Comparator: Conventional Lecture Program

#### Randomization:

• Individual-level randomization using simple randomization (computer-generated list).

### 5. Study Population

Participants: Fifth-semester nursing students.

Inclusion Criteria:

- Registered in the targeted semester and course.
- Provide informed consent.

## **Exclusion Criteria:**

- Prior exposure to VR dementia training.
- Not enrolled in designated courses.

#### 6. Recruitment Procedures

Recruitment through class announcement, LMS, and Google Forms.

Participants assigned new unique IDs to protect confidentiality.

Study explained via Zoom (control group) and in class (intervention group).

### 7. Interventions

Experimental Arm (VR Program):

- Single-session VR dementia education program with max 20 students.
- Components include introduction, questionnaires, undesirable and desirable VR, dramas, lectures, N-impro, reflection, and conclusion.

#### Control Arm:

- Study briefing + pre-test via Zoom.
- Conventional dementia lecture via LMS.
- Post-test via Zoom.
- Summary assignment required.

#### 8. Outcome Measures

### Primary Outcome:

• Attitudes Toward People With Dementia Scale (14 items).

## Secondary Outcomes:

- Dementia Knowledge Scale
- Intention to Help (vignettes)
- User Experience Questionnaire (UEQ) for intervention arm

# 9. Statistical Analysis Plan (SAP)

**Analysis Principles:** 

- Intention-to-treat (ITT) analysis.
- Significance level:  $\alpha = 0.05$  (two-sided).
- Missing data handled by multiple imputation if >5%.

## Primary Outcome Analysis:

- Compare change in attitude scores (T1 to T2 and T1 to T3) between groups.
- Independent t-test or Mann–Whitney U (non-parametric).
- Repeated-measures ANOVA or mixed-effects model for time × group interaction.

### Secondary Outcomes:

- Knowledge: Pre-post difference tested using paired t-test, ANCOVA controlling baseline.
- Intention to help: Likert-scale comparisons using Mann-Whitney U.
- UEQ: Descriptive statistics, domain scores, and comparison with normative database.

## Subgroup Analyses:

- Gender
- Prior dementia experience (family exposure)

## Sample Size:

• Estimated 60 intervention, 150 control (educational-program constraints).

## Data Monitoring:

• Conducted internally by the research team.

### Software:

SPSS 29 / R version 4.3

10. Ethical Considerations

Ethics approval: KEPK 3922-KEPK.

Confidentiality protected through new unique participant IDs.

Participation voluntary; withdrawal allowed at any time.

## Data Storage:

• Encrypted drive, stored for 5 years, accessible only to PI and research team.

11. Timeline

Recruitment: Sept—Oct 2025
Intervention: Oct—Nov 2025
Follow-up: Jan—Feb 2026

• Analysis & Reporting: Mar-May 2026

## References

- 1. Jhang KM, Chang MC, Lo TY, Lin CW, Wang WF, Wu HH. Using the apriori algorithm to classify the care needs of patients with different types of dementia. Patient Prefer Adherence. Dove Medical Press Ltd.; 2019;13:1899–912.
- 2. Merrill MD. First Principles of Instruction. WTR&D. 2002;50:43-59.
- 3. Vanderbilt C and TG at. The Jasper experiment: An exploration of issues in learning and instructional design. Educational Technology Research and Development. 1992;40:65–80.
- 4. Phillipson L, Hall D, Cridland E, Fleming R, Brennan-Horley C, Guggisberg N, et al. Involvement of people with dementia in raising awareness and changing attitudes in a dementia friendly community pilot project. Dementia. SAGE Publications Ltd; 2019;18:2679–94.
- 5. Gilmartin-Thomas JFM, McNeil J, Powell A, Malone DT, Wolfe R, Larson IC, et al. Impact of a Virtual Dementia Experience on Medical and Pharmacy Students' Knowledge and Attitudes Toward People with Dementia: A Controlled Study. Journal of Alzheimer's Disease. IOS Press; 2018:62:867–76.
- 6. Matsumoto H, Igarashi A, Sakka M, Takaoka M, Kugai H, Ito K, et al. A Two-Step Model for Encouraging the General Public to Exhibit Helping Behaviors Toward People Living with Dementia. Innov Aging. Oxford University Press; 2022;6.
- 7. Sari DW, Igarashi A, Takaoka M, Yamahana R, Chie MN, Yamamoto-mitani N. Virtual reality program to develop dementia-friendly communities in Japan. Australas J Ageing [Internet]. 2020;39:1–8. Available from: <a href="https://onlinelibrary.wiley.com/doi/10.1111/ajag.12797">https://onlinelibrary.wiley.com/doi/10.1111/ajag.12797</a>
- 8. Suzuki H, Igarashi A, Yamamoto-Mitani N. Effects of a dementia educational program using virtual reality on the attitude of general public toward people living with dementia: A randomized controlled trial. 2023.

- 9. Wu, J., Igarashi, A., Suzuki, H., Matsumoto, H., Kugai, H., Takaoka, M., & Yamamoto-Mitani, N. (2024). Effects of a dementia educational programme using virtual reality on nurses in an acute care hospital: A pre-post comparative study. International Journal of Older People Nursing, 19, e12616. https://doi.org/10.1111/opn.12616Igarashi A, Matsumoto H, Takaoka M, Kugai H, Suzuki M, Yamamoto-Mitani N. Educational Program for Promoting Collaboration Between Community Care Professionals and Convenience Stores. Journal of Applied Gerontology. SAGE Publications Inc.; 2020;39:760–9.
- 10. Igarashi A, Matsumoto H, Takaoka M, Kugai H, Suzuki M, Yamamoto-Mitani N. Educational program for promoting collaboration between community care professionals and convenience stores in Japan. Journal of Applied Gerontology. 2019;1–20.
- 11. Matsumoto H, Hagiwara Y, Yamamoto-Mitani N, Igarashi A. A randomized control trial for ReDeSign: A dementia- friendly mobile microlearning training for store workers in Japan. Gerontologist. 2022;1–22.
- 12. Matsumoto H, Igarashi A, Suzuki M, Yamamoto-Mitani N. Association between neighbourhood convenience stores and independent living in older people in Japan. Australas J Ageing. 2019;38:116–23.
- 13. Igarashi A, Matsumoto H, Suzuki M, Aoki S, Aburayama K, Murata S, et al. Use of convenience stores in community- dwelling older adults who utilize home help services offered under the long-term care insurance: A cross-sectional questionnaire survey for older adult cases that convenience store provides support in daily life. Japan Socio-Gerontological Society. 2018;40:283–91.
- 14. Igarashi A, Eltaybani S, Takaoka M, Noguchi-Watanabe M, Yamamoto-Mitani N. Quality Assurance in Long-Term Care and Development of Quality Indicators in Japan. Gerontol Geriatr Med. 2020;6.
- 15. Aihara Y, Maeda K. National dementia supporter programme in Japan. Dementia. SAGE Publications Ltd; 2021;20:1723–8.
- 16. World Health Organization. Towards age-friendly primary health care. World Health Organization; 2004.
- 17. Leroi I, Kitagawa K, Vatter S, Sugihara T. Dementia in 'super-aged' Japan: challenges and solutions. Neurodegener Dis Manag. 2018;8.
- 18. Ministry of Foreign Affairs of Japan. Japan-Indonesia Economic Partnership Agreement [Internet]. 2022. Available from: <a href="https://www.mofa.go.jp/policy/economy/fta/indonesia.html">https://www.mofa.go.jp/policy/economy/fta/indonesia.html</a>
- 19. World Health Organization. Risk reduction of cognitive decline and dementia WHO guidelines. 2020.
- 20. Freel S. The Global Dementia Observatory Reference Guide World Health Organization [Internet]. 2018. Available from: <a href="http://apps.who.int/bookorders">http://apps.who.int/bookorders</a>.
- 21. Global action plan on the public health response to dementia [Internet]. Available from: <a href="http://apps.who.int/bookorders">http://apps.who.int/bookorders</a>.
- 22. Ministry of health L and WJ. Comprehensive Strategy for Promotion of Dementia Measures-Towards Community Development Friendly to Elderly People with Dementia-(New Orange Plan) [Internet]. 2015 [cited 2023 Apr 24]. Available from: <a href="https://www.mhlw.go.jp/stf/houdou/000072246.html">https://www.mhlw.go.jp/stf/houdou/0000072246.html</a>
- 23. Awata S. [Medical services for dementia in the Comprehensive Strategy to Accelerate Dementia Measures (New Orange Plan)]. Nihon Rinsho [Internet]. 2016 [cited 2023 Apr 24];74:499–504. Available from: <a href="https://pubmed.ncbi.nlm.nih.gov/27025094/">https://pubmed.ncbi.nlm.nih.gov/27025094/</a>

- 24. Hebditch M, Daley S, Wright J, Sherlock G, Scott J, Banerjee S. Preferences of nursing and medical students for working with older adults and people with dementia: A systematic review. BMC Med Educ. BioMed Central Ltd.; 2020;20.
- 25. Japan Association of Colleges of Nursing. Core Competencies and Goals for Achievement at Graduation in Bachelor's Degree Nursing Education [Internet]. Available from: https://doi.org/10.32283/rep.5618b431
- 26. Giuseppe R. Virtual Reality. Encyclopedia of Biomedical Engineering. Wiley & Sons, Inc.; 2006;1–17.
- 27. Dyer E, Swartzlander BJ, Gugliucci MR. Using virtual reality in medical education to teach empathy. Journal of the Medical Library Association. 2018;106:498–500.
- 28. Adefila A, Graham S, Clouder L, Bluteau P, Ball S. myShoes the future of experiential dementia training? Journal of Mental Health Training, Education and Practice. Emerald Group Publishing Ltd.; 2016;11:91–101.
- 29. Hirt J, Beer T. Use and impact of virtual reality simulation in dementia care education: A scoping review. Nurse Educ Today. Churchill Livingstone; 2020.
- 30. Suzuki H, Igarashi A, Sakai S, Sakka M, Takaoka M, Matsumoto H, et al. Effectiveness of a dementia educational program to provide a first-person experience on the attitude of nursing students toward people living with dementia: A prospective observational study. Journal of Japanese Society for Dementia Care 22 (2), 393-403, 2023Kim K, Kuroda K. Factors related to attitudes toward people with dementia: Development Attitude Toward Dementia Scale and Dementia Knowledge Scale. Bulletin of Social Medicine. 2011;28:43-56 (in Japanese).
- 31. Bibb L, Darley JM. The unresponsive bystander: why doesn't he help? . Appleton-Century Crofts; 1970.
- 32. Mikami M, Nakao R, Horikawa R, Sugiyama K, Sawada Y, Kirino M, et al. Developing a scale to assess dementia- related knowledge among local residents. Bulletin of Social Medicine. 2017;18:30.
- 33. Matsumoto H, Igarashi A, Suzuki M, Mitani N. Association between neighbourhood convenience stores and independent living in older people in Japan. Australasian Journal of Ageing

# INFORMED CONSENT FORM

Dear participant,

We invite nursing students to complete the questionnaire below.

Information about this study:

Title : The Effect of a Comprehensive Dementia Education Program on

Improving Attitudes Toward People Living with Dementia: A

Randomized Controlled Trial

Purpose : To identify the effect of a Comprehensive Dementia Education

Program on improving nursing students' attitudes toward people living

with dementia.

Principal Investigator: Dianis Wulan Sari, Faculty of Nursing, Universitas Airlangga

Contact Person : Dianis; 0812-5949-7373

Study Period : October 1, 2025 – May 30, 2026

This study is administered once and will take about 90 minutes.

We would like to assure you that:

- Your participation in this study is voluntary. You have the right to refuse or agree to participate.
- Your information will be treated anonymously and confidentially, and will not be used for purposes other than this research.
- You may leave questions unanswered without penalty.
- Your responses will be stored in an encrypted drive and will be deleted five years after the publication of the research.

Completing and returning this questionnaire signifies your consent to participate in this study. Once your response is submitted, it cannot be withdrawn.

| Do you agree to participate in this survey? |
|---------------------------------------------|
| □ Yes, I agree |
| □ No, I do not agree |

This statement is made to be used as necessary.